CLINICAL TRIAL: NCT01268423
Title: Impact of Early Percutaneous Tracheostomy on the Incidence of Swallowing Dysfunction in Critically Ill Patients on Mechanical Ventilation. A Randomized Clinical Trial
Brief Title: Early Percutaneous Tracheostomy and Swallowing Dysfunction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Carlos Romero. Principal Investigator, Universidad de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FONIS SA10I20012
Record Dates: First submitted 2010-12-29; First posted 2010-12-30 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2010-12

CONDITIONS: Swallowing Disorder
Keywords: Percutaneous tracheostomy; Swallowing dysfunction; Mechanical ventilation; Intensive Care
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early percutaneous tracheostomy (Experimental)
  Interventions: Procedure: Percutaneous tracheostomy
- Prolonged translaryngeal intubation (Active Comparator)
  Interventions: Procedure: Prolonged translaryngeal intubation

INTERVENTIONS:
Procedure: Percutaneous tracheostomy — Percutaneous tracheostomy within the first 4 days of mechanical ventilation.
  Other Names: Percutaneous dilatational tracheostomy
  Arms: Early percutaneous tracheostomy
Procedure: Prolonged translaryngeal intubation — Prolonged endotracheal intubation, and reevaluation at day 10 to establish the requirement of percutaneous tracheostomy. If clinical condition determines that the patient needs a percutaneous tracheostomy, this will be performed between days 11 and 14.
  Other Names: Prolonged endotracheal intubation
  Arms: Prolonged translaryngeal intubation

SUMMARY:
The aim of the study is to determine if performing an early tracheostomy (within the first 4 days of endotracheal intubation) in critically ill patients on mechanical ventilation, reduces the incidence of swallowing dysfunction.

DETAILED DESCRIPTION:
The development of initial resuscitation maneuvers, associated with a better knowledge of the physiopathology of critical illnesses and the technological development experienced by critical care medicine, allow us to give vital support to patients for long periods of time. In this scenario, a considerable proportion of critically ill patients may require translaryngeal intubation and invasive mechanical ventilation. Patients who require prolonged translaryngeal intubation have a high risk of developing swallowing dysfunction, a condition predisposing to secretions aspiration. Until now, there has been no demonstration of a causal association between the duration of translaryngeal intubation and development of swallowing dysfunction. However, all the studies about this topic have been performed on patients submitted to prolonged translaryngeal intubation. Clinical studies have documented the development of early laryngotracheal lesions after intubation, which might explain post extubation dysfunction of swallowing reflex, probably as consequence of alteration of mechanic and chemo-receptors of the pharyngeal and laryngeal mucosa. There are no studies evaluating the impact of an early percutaneous tracheostomy on the incidence of swallowing dysfunction in critical care patients. The investigators have documented a 38% of swallowing dysfunction in our critically ill patients submitted to prolonged mechanical ventilation. The hypothesis of the study is that performance of an early percutaneous tracheostomy, within the first 4 days of translaryngeal intubation, in critical care patients on mechanical ventilation, reduces the incidence of swallowing dysfunction. The diagnosis of swallowing dysfunction will be performed by fiberoptic endoscopic evaluation of swallowing (FEES) by a trained otolaryngologist, 3 to 5 days after weaning of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained for the procedure
* Patients whose need of mechanical ventilation is estimated in ≥ 7 days and require a percutaneous tracheostomy

Exclusion Criteria:

* Patients younger than 18 years old
* Patients with neurologic pathology
* Patients with dysphagia history
* Patients whose MV duration is estimated in < 7 days
* Patients with airway obstruction requiring an emergency tracheostomy
* Patients already having a tracheostomy in situ
* Pregnancy
* Patients who have already been enrolled on another trial
* Patients with absolute contraindication to perform a percutaneous tracheostomy
* Patients with high risk of dying, life expectancy of < 48 hours
* Patients in whom limitation of therapy has been decided
* Family rejection to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of swallowing dysfunction | 3 to 5 days after weaning of mechanical ventilation
  The diagnosis of swallowing dysfunction will be performed by fiberoptic endoscopic evaluation of swallowing (FEES) 3 to 5 days after weaning of mechanical ventilation.

SECONDARY OUTCOMES:
Ventilator-free days | 28 days
Incidence of ventilator-associated pneumonia | 28 days
Delirium-free and coma-free days | 28 days
Daily dose of sedatives | 28 days
ICU-free days | 28 days
Critical Care Unit-free days | 90 days
  Length of stay at Critical Care Unit involve days of stay in thre Intensive Care Unit, plus the days of stay in the Intermediate Care Unit.
Hospital length of stay | 90 days
All cause mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Romero, MD, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile